CLINICAL TRIAL: NCT05533008
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Potential of Physical Withdrawal From Intravenous CR845 (Difelikefalin) in Hemodialysis Patients
Brief Title: CR845-100303: Study to Assess the Potential of Physical Withdrawal From Intravenous CR845 (Difelikefalin) in Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR845-100303
Record Dates: First submitted 2019-11-19; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Hemodialysis
Keywords: Difelikefalin; CR845; Physical Withdrawal; Hemodialysis; Dialysis; CKD; ESRD (end stage renal disease); Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CR845 0.5 mcg/kg (Experimental): IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 0.5 mcg/kg
- Placebo (Placebo Comparator): IV Placebo administered after each dialysis session (3 times/week)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg — IV CR845 0.5 mcg/kg as a bolus injection
  Other Names: Difelikefalin
  Arms: CR845 0.5 mcg/kg
Other: Placebo — IV Placebo as a bolus injection
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to assess the potential of physical withdrawal from CR845 upon treatment discontinuation after 3 weeks of IV administration at a dose of 0.5 mcg/kg in hemodialysis patients. The purpose of this study is to determine whether hemodialysis patients who take CR845 develop physical dependence and experience withdrawal symptoms upon cessation, as exemplified by symptoms consistent with opioid withdrawal. The study will consist of a Screening Phase, a 3-week Open-label Phase, a 2-week randomized, placebo-controlled, Double-blind Phase and a Follow-up Visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Has ESRD and has been on hemodialysis 3 times per week for at least 3 months;
* Not currently taking opioid medication;
* If female, is not pregnant or nursing during any period of the study.

Key Exclusion Criteria:

• Has a concomitant disease or a history of any condition that, in the opinion of the Investigator, could pose undue risk to the patient, impede completion of the study procedures, or would compromise the validity of the study measurements; Past or present diseases, which as judged by the Investigator, may affect the outcome of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Treatment difference between placebo and CR845-treated group with respect to the maximum Clinical Opiate Withdrawal Scale (COWS) score over Weeks 1-4 | Week 1-4

SECONDARY OUTCOMES:
Treatment difference between placebo and CR845-treated group for COWS score at Week 4. | Week 4
Treatment difference between placebo and CR845-treated group for COWS score at Week 5. | Week 5
Treatment difference between placebo and CR845-treated group for maximum Subjective Opiate Withdrawal Scale (SOWS) score over Weeks 1-4 | Week 1-4
Treatment difference between placebo and CR845-treated group for SOWS score at Week 4. | Week 4
Treatment difference between placebo and CR845-treated group for SOWS score at Week 5. | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (5):
- United States (5):
  - Cara Therapeutics Study Site, Bridgeport, Connecticut
  - Cara Therapeutics Study Site, Hartford, Connecticut
  - Cara Therapeutics Study Site, Kansas City, Kansas
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No